CLINICAL TRIAL: NCT03004989
Title: Experiences of Participating in Return to Work Group Programmes for People With Musculoskeletal Disorders: A Focus Group Study
Brief Title: Experiences of Participating in Return to Work Group Programmes
Acronym: RTW-GP
Status: Completed | Type: Observational
Sponsor: Revmatismesykehuset AS (Other)
Collaborators: South-Eastern Norway Regional Health Authority (Other)
Responsible Party: Sponsor
Other Study IDs: 2012/7266 UiO
Record Dates: First submitted 2016-12-20; First posted 2016-12-29 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-12

CONDITIONS: Musculoskeletal Diseases or Conditions
Keywords: Qualitative study; Musculoskeletal Disorders; Return to Work Programme
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Programme 1: RTW group in day clinics
  Interventions: Behavioral: Programme
- Programme 2: RTW group in day clinics for people with fibromyalgia
  Interventions: Behavioral: Programme
- Programme 3: My work and I
  Interventions: Behavioral: Programme

INTERVENTIONS:
Behavioral: Programme — The participants of this study had participated in one of three different RTW-GPs. These programmes are designed to enable participants to proactively take action in their daily lives and in collaboration with employers achieve the best possible working conditions. All the group sessions are based on cognitive theory where attention, awareness and reflection on one's own work and life situation is important
  Other Names: Programme 1; Programme 2; Programme 3

SUMMARY:
To explore the experiences of individuals with musculoskeletal disorders (MSDs) who have participated in return-to-work group programmes (RTW-GPs) and see how the programmes could strengthen their work ability.

DETAILED DESCRIPTION:
For a representative sampling of experiences, participants who had participated in various groups over time in outpatient and inpatient groups in the RTW-GP were invited to enrol in the study. Other inclusion criteria were age between 25 and 65 years, different musculoskeletal diagnosis and that they should come from the rural district/city of residence.

The participants received requests by letter to participate in the focus group interview six months after the final group intervention, the same time as they were invited to a follow-up visit. Only a few men had participated in the RTW-GPs and none of them wanted to take part in the study.

All participants were given written and oral information about the study, the use of recording and transcribing devices, and their right to withdraw from the study at any time. The interviews were carried out after the participants gave written, informed consent.

Three focus group interviews were conducted: one with six participants, and two with five. One participant who could not participate in the focus group interview participated at an individual interview with the same questions as in the focus groups. The individual interview was conducted first and served as a test for the questions in the interview guide.

Interventions The participants of this study had participated in one of three different RTW-GPs. These programmes are designed to enable participants to proactively take action in their daily lives and in collaboration with employers achieve the best possible working conditions. All the group sessions are based on cognitive theory where attention, awareness and reflection on one's own work and life situation is important. Motivation is instilled by helping participants recognise opportunities for change. Participants set work-related goals and receive individual feedback from multidisciplinary personnel in addition to various group-based sessions with teaching, activities and exercises. The participants are referred to the programme by a rheumatologist or a member of the hospital's multidisciplinary team as soon as possible after starting sick-leave.

ELIGIBILITY:
Inclusion Criteria:

* Participating RTW-GP
* Musculoskeletal diagnoses
* From the rural district/city of residence
* Speaking Norwegian

Ages: 28 Years to 57 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: A total of 17 female informants participated in the study, age 28 - 57 years
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2012-05; Primary Completion 2013-11 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Patient experiences after participating at RTW-GP | May 2012 - November 2013
  Focus group interviews
Quality of life | May 2012 - November 2013
  Focus group interviews
Work ability | May 2012 - November 2013
  Focus group interview

CONTACTS AND LOCATIONS:
Overall Officials: Bente Hamnes, PhD, Study Chair — Revmatismesykehuset AS
Locations (1):
- Revmatismesykehuset, Lillehammer, Norway

IPD SHARING:
Plan to Share IPD: No